CLINICAL TRIAL: NCT06582615
Title: Food for Thought - Pilot Study of a MIND Diet Intervention in Women Undergoing Active Treatment for Triple Negative Breast Cancer
Brief Title: Food for Thought - A Nutrition Intervention for Women Undergoing Active Treatment for Triple Negative Breast Cancer
Acronym: MIND-TNBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Tonya Orchard, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-23384; NCI-2024-05451 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Specimen Handling; Mental Status and Dementia Tests; Diet Therapy

STUDY DESIGN:
Intervention Model Description: Parallel design with optional cross-over of the control group to the treatment group after 6-month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (MIND-TNBC counseling) (Experimental): Patients receive MIND counseling sessions over 30-60 minutes weekly for 4 weeks then over 15 minutes biweekly for 4 sessions over 8 weeks and follow a personalized diet for 12 weeks. Patients also wear a Fitbit and undergo dried blood spot collection on study and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Other: Dietary Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration
- Arm II (general health recommendations counseling) (Active Comparator): Patients receive general health recommendations counseling sessions over 30-60 minutes weekly for 4 weeks then over 15 minutes biweekly for 4 sessions over 8 weeks. Patients also wear a Fitbit and undergo dried blood spot collection on study and during follow up. After 6 month follow-up, patients may receive the MIND counseling sessions as in Arm I.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Other: Dietary Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo dried blood spot collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cognitive Assessment — Ancillary studies
Other: Dietary Intervention — Receive MIND counseling sessions
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (MIND-TNBC counseling)
Other: Dietary Intervention — Follow a personalized diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (MIND-TNBC counseling)
Other: Dietary Intervention — Receive general health recommendations counseling sessions
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm II (general health recommendations counseling)
Other: Medical Device Usage and Evaluation — Wear a Fitbit
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The goal of this randomized clinical trial is to learn if a healthy eating pattern called the MIND eating plan can reduce cancer-related cognitive impairment (commonly called "chemobrain") and other symptoms commonly experienced by women with newly diagnosed stage II-III triple negative breast cancer as they go through chemotherapy. The symptoms that will be measured include changes in memory and mental function, fatigue, sleep quality, anxiety, and depression.

Researchers will compare measures from women in the 12-week MIND eating plan virtual intervention to a general health coaching (GHC) virtual intervention to see if the MIND eating plan helps reduce symptoms. Women will be contacted for follow-up measures 6 months after the 12-week interventions.

Women randomly assigned to the GHC at the beginning of the study will have the opportunity to complete the MIND intervention after the 6-month follow-up. All study sessions and measures are done remotely.

Participants will:

* Be randomized to MIND or GHC interventions
* Complete all study measures remotely (by online questionnaires, virtual visits and mail )
* Attend 8 virtual sessions of about 15-60 minutes each over 12 weeks
* Be sent some of the key foods in the MIND eating plan during the MIND intervention
* Be contacted for follow-up measures 6 months after interventions

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the efficacy of a remotely delivered, highly accessible, 3-month MIND diet intervention (MIND-Breast Cancer [BC]) versus (vs.) general health curriculum (GHC) control to reduce CRCI and associated neuropsychological symptoms in 60 racially and ethnically diverse women with clinical stage II-III TNBC.

II. Evaluate the sustainability of dietary changes and outcome measures 6-months post-intervention.

EXPLORATORY OBJECTIVE:

I. Explore underlying mechanisms of the MIND-BC diet on CRCI and effects of early versus later participation in the dietary intervention.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive MIND counseling sessions over 30-60 minutes weekly for 4 weeks then over 15 minutes biweekly for 4 sessions over 8 weeks and follow a personalized diet for 12 weeks. Patients also wear a Fitbit and undergo dried blood spot collection on study and during follow up.

ARM II: Patients receive general health recommendations counseling sessions over 30-60 minutes weekly for 4 weeks then over 15 minutes biweekly for 4 sessions over 8 weeks. Patients also wear a Fitbit and undergo dried blood spot collection on study and during follow up. After 6 month follow-up, patients may receive the MIND counseling sessions as in Arm I.

After completion of study intervention, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years
* Female with stage I-III triple negative breast cancer
* Less than or equal to 12 months from starting initial systemic cancer treatment (e.g. chemotherapy, targeted therapy, immunotherapy) for TNBC
* Ability to access and use internet resources, including video calls using Zoom platform
* English speaking

Exclusion Criteria:

* History of dementia, stroke, traumatic brain injury, brain metastasis or other conditions that could lead to cognitive impairment
* Current healthy eating pattern reflected by high MIND diet score (e.g. >12)
* Unwilling/unable to eat > 2 types of MIND food (e.g. avoids & > 2 categories or food groups such as leafy greens, olive oil and non-fried fish)
* Currently pregnant
* Unable to give informed consent

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Wechsler Adult Intelligence Scale, fourth edition (WAIS-IV) Digit Span score | Baseline up to 6 months post-intervention
  Analyses of change in WAIS-IV test scores will be based on a linear or generalized linear mixed effects regression model, as appropriate. Timepoint, treatment assignment, and their interaction will be included as fixed effects, and a subject-level random intercept effect will be included to account for correlation of repeated measurements from the same subject. Pathological complete response and baseline measurements of the outcome variables will also be included as fixed effects to improve precision, as will any demographic variables that are substantially imbalanced at baseline. Will report descriptive statistics, and when applicable, comparisons between randomized groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Orchard, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu